CLINICAL TRIAL: NCT05882877
Title: A Phase 3, Multicenter, Double-blind Maintenance Study to Assess Long-term Safety, Tolerability, and Efficacy of Rocatinlimab in Adult and Adolescent Subjects With Moderate-to-severe Atopic Dermatitis (AD) (ROCKET-ASCEND)
Brief Title: A Study to Assess Long-term Safety, Tolerability, and Efficacy of Rocatinlimab in Adult and Adolescent Participants With Moderate-to-severe Atopic Dermatitis (AD)
Acronym: ROCKET-ASCEND
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20210146; 2022-501587-17 (EudraCT Number)
Record Dates: First submitted 2023-05-22; First posted 2023-05-31 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Rocatinlimab; AMG 451; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — KHK4083

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- ARM A: Dose 1 to Dose 1 (Experimental): Participants from parent Rocatinlimab studies ROCKET-Ignite, ROCKET-Horizon, ROCKET-SHUTTLE, or ROCKET-ASTRO who received Dose 1 will be randomized or assigned to receive Dose 1 Every 4 Weeks (Q4W) or Every 8 Weeks (Q8W). Participants from parent Rocatinlimab study ROCKET-VOYAGER who received Dose 1 will be assigned to receive Dose 1 Q4W.
  Interventions: Drug: Rocatinlimab
- ARM B: Dose 2 to Dose 2 (Experimental): Participants from parent Rocatinlimab studies ROCKET-Ignite, ROCKET-SHUTTLE, or ROCKET-ASTRO who received Dose 2 will be randomized or assigned to receive Dose 2 Q4W or Q8W.
  Interventions: Drug: Rocatinlimab
- ARM C: Dose 1 or Dose 2 to Placebo (Placebo Comparator): Participants from parent Rocatinlimab studies ROCKET-Ignite or ROCKET-Horizon who received Dose 1 will be randomized to receive placebo Q4W. Participants from parent Rocatinlimab study ROCKET-Ignite who received Dose 2 will be randomized to receive placebo Q4W.
  Interventions: Other: Placebo
- ARM D: Placebo to Placebo (Placebo Comparator): Participants from parent Rocatinlimab studies ROCKET- Ignite, ROCKET-Horizon, ROCKET-SHUTTLE, ROCKET-ASTRO, or ROCKET-VOYAGER who received placebo will be randomized or assigned to receive placebo Q4W.
  Interventions: Other: Placebo
- ARM E: Dose 1, Dose 2, Placebo, or Open-label (OL) to OL Dose 1 (Experimental): Participants from parent Rocatinlimab studies ROCKET- Ignite, ROCKET-Horizon, ROCKET- SHUTTLE, ROCKET-ASTRO, or ROCKET-VOYAGER who received Dose 1, Dose 2, or placebo will be assigned to receive OL Rocatinlimab Dose 1 Q4W.
  Participants who received OL in parent Rocatinlimab study ROCKET- ASTRO will continue to receive OL Rocatinlimab Dose 1 Q4W.
  All participants from parent Rocatinlimab study ROCKET-Orbit will continue to receive OL Rocatinlimab Dose 1 Q4W.
  Interventions: Drug: Rocatinlimab
- ARM F Group (No Intervention): Participants in Arm E (OL Rocatinlimab Dose 1 Q4W) who meet defined criteria will have Rocatinlimab withdrawn, but will continue all subsequent study visits.
- ARM G Group (Experimental): Participants from Arm F who meet defined criteria will resume OL Rocatinlimab Dose 1 Q4W.
  Interventions: Drug: Rocatinlimab

INTERVENTIONS:
Drug: Rocatinlimab — Subcutaneous (SC) injection
  Other Names: AMG 451; KHK4083
  Arms: ARM A: Dose 1 to Dose 1; ARM B: Dose 2 to Dose 2; ARM E: Dose 1, Dose 2, Placebo, or Open-label (OL) to OL Dose 1; ARM G Group
Other: Placebo — SC injection
  Arms: ARM C: Dose 1 or Dose 2 to Placebo; ARM D: Placebo to Placebo

SUMMARY:
The primary objective of this study is to describe the long-term safety and tolerability of rocatinlimab in participants with moderate-to-severe AD.

ELIGIBILITY:
Inclusion Criteria:

* Completion of an end of treatment duration visit (Week 24 or Week 52 visit for adult or adolescent studies, respectively) in a rocatinlimab parent study (ROCKET-IGNITE, ROCKET-HORIZON, ROCKET-SHUTTLE, ROCKET-ASTRO, ROCKET-ORBIT, OR ROCKET-VOYAGER) within the past 28 days.
* Participants from the parent study ROCKET-ORBIT must achieve an improvement in EASI score at week 52 of at least 60% compared to parent study baseline (EASI 60).

Exclusion Criteria:

* Permanent investigational product discontinuation due to safety-related reasons, protocol-defined stopping rules or conditions/reasons unrelated to efficacy during the rocatinlimab parent study (ROCKET-IGNITE, ROCKET-HORIZON, ROCKET-SHUTTLE, ROCKET-ASTRO, ROCKET-ORBIT, OR ROCKET-VOYAGER), or at the time of Screening or Day 1.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2621 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events | Up to 116 weeks

SECONDARY OUTCOMES:
Maintaining Validated Investigator's Global Assessment for Atopic Dermatitis (vIGA-AD™) 0/1 Response at Week 32 Among Participants Achieving vIGA-AD™ 0/1 Response at Day 1 | Week 32
  This outcome measure applies only to participants from parent rocatinlimab studies ROCKET-Ignite and ROCKET-Horizon who entered into the randomized treatment withdrawal cohort.
Maintaining a Revised IGA (rIGA™) 0/1 Response at Week 32 Among Participants Achieving rIGA™ 0/1 Response at Day 1 | Week 32
  This outcome measure applies only to participants from parent rocatinlimab studies ROCKET-Ignite and ROCKET-Horizon who entered into the randomized treatment withdrawal cohort.
Maintaining Eczema Area and Severity Index (EASI) 75 Response at Week 32 Among Participants Achieving EASI 75 Response at Day 1 | Week 32
  This outcome measure applies only to participants from parent rocatinlimab studies ROCKET-Ignite and ROCKET-Horizon who entered into the randomized treatment withdrawal cohort.
Maintaining EASI 90 Response at Week 32 Among Participants Achieving EASI 90 Response at Day 1 | Week 32
  This outcome measure applies only to participants from parent rocatinlimab studies ROCKET-Ignite and ROCKET-Horizon who entered into the randomized treatment withdrawal cohort.
Maintaining vIGA-AD™ 0/1 Response and EASI 75 Response at Week 32 Among Participants Achieving vIGA-AD™ 0/1 Response and EASI 75 Response at Day 1 | Week 32
  This outcome measure applies only to participants from parent rocatinlimab studies ROCKET-Ignite and ROCKET-Horizon who entered into the randomized treatment withdrawal cohort.
Maintaining ≥ 4-point Reduction from Parent Study Baseline in Worst Pruritus NRS Score at Week 32 Among Participants Achieving ≥ 4 Point Reduction from Parent Study Baseline in Worst Pruritus NRS Score at Day 1 | Week 32
  This outcome measure applies only to participants from parent rocatinlimab studies ROCKET-Ignite and ROCKET-Horizon who entered into the randomized treatment withdrawal cohort.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (547):
- United States (136):
  - Cahaba Dermatology and Skin Health Center, Birmingham, Alabama
  - Medical Dermatology Specialists, Phoenix, Arizona
  - Alliance Dermatology and Mohs Center, Phoenix, Arizona
  - Affiliated Dermatology, Scottsdale, Arizona
  - Scottsdale Clinical Trials, Scottsdale, Arizona
  - Dermatology Trial Associates, Bryant, Arkansas
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Arkansas Research Trials, LLC, North Little Rock, Arkansas
  - Kern Research Inc, Bakersfield, California
  - Hope Clinical Research LLC, Canoga Park, California
  - West Coast Research LLC, Dublin, California
  - California Dermatology and Clinical Research Institute, Encinitas, California
  - First OC Dermatology, Fountain Valley, California
  - Antelope Valley Clinical Trials, Lancaster, California
  - Chemidox Clinical Trials Incorporated, Lancaster, California
  - Long Beach Research Institute, Long Beach, California
  - University of California Los Angeles, Los Angeles, California
  - Dermatology Research Associates, Los Angeles, California
  - Wallace Medical Group Inc, Los Angeles, California
  - Northridge Clinical Trials, Northridge, California
  - University of California Irvine, Orange, California
  - Havana Research Institute Inc, Pasadena, California
  - Integrative Skin Science and Research, Sacramento, California
  - University of California at Davis Medical Center, Sacramento, California
  - Kaiser Permanente South Sacramento Medical Center, Sacramento, California
  - Alliance Clinical Research, San Diego, California
  - Kaiser Permanente Medical Center - Oakland, San Francisco, California
  - Kaiser Permanente Medical Center - San Francisco, San Francisco, California
  - Wolverine Clinical Trials, Santa Ana, California
  - Clinical Science Institute, Santa Monica, California
  - IMMUNOe Research Centers, Centennial, Colorado
  - Skin Care Research Incorporated, Boca Raton, Florida
  - Renaissance Research and Medical Group, Cape Coral, Florida
  - Driven Research LLC, Coral Gables, Florida
  - Corazon United States of America, LLC doing business as Life Clinical Trials, Coral Springs, Florida
  - D and H Doral Research Centers, Doral, Florida
  - Saint Jude Clinical Research, Doral, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Global Research Solutions, Homestead, Florida
  - Nexus Clinical Research, Homestead, Florida
  - Glick Skin Institute, Margate, Florida
  - ara Professionals Limited Liability Corporation, Miami, Florida
  - Gold Coast Health Research Center, Miami, Florida
  - Miami Clinical Research, Miami, Florida
  - Healthy Life Research, Miami, Florida
  - Anchor Medical Research, Miami, Florida
  - Meridian International Research, Miami Gardens, Florida
  - Savin Medical Group LLC, Miami Lakes, Florida
  - Clinical Associates of Orlando Limited Liability Company, Orlando, Florida
  - Innovation Medical Research Center Inc, Palmetto Bay, Florida
  - University of South Florida, Tampa, Florida
  - Olympian Clinical Research - Tampa, Tampa, Florida
  - Atlanta Dermatology, Vein and Research Center, PC, Alpharetta, Georgia
  - First Georgia Physicians Group, Fayetteville, Georgia
  - Advanced Medical Research PC, Sandy Springs, Georgia
  - Treasure Valley Medical Research, Boise, Idaho
  - DeNova Research, Chicago, Illinois
  - Sneeze, Wheeze, and Itch Associates, LLC, Normal, Illinois
  - Endeavor Health Clinical Trials Center, Skokie, Illinois
  - Dundee Dermatology, West Dundee, Illinois
  - DS Research, Clarksville, Indiana
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Southern Indiana Clinical Trials, New Albany, Indiana
  - The Indiana Clinical Trials Center PC, Plainfield, Indiana
  - Options Research Group LLC, West Lafayette, Indiana
  - Dermatology and Skin Cancer Center Leawood, Leawood, Kansas
  - DS Research, Louisville, Kentucky
  - Kentucky Advanced Medical Research LLC, Murray, Kentucky
  - Foxhall Research Center, Chevy Chase, Maryland
  - Institute for Asthma and Allergy, Chevy Chase, Maryland
  - Continental Clinical Solutions, LLC, Towson, Maryland
  - MetroBoston Clinical Partners, Brighton, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Medical Center - New Center One, Detroit, Michigan
  - Onyx Clinical Research, Flint, Michigan
  - Revival Research Institute LLC, Troy, Michigan
  - Somerset Skin Centre, Troy, Michigan
  - Dermatology and Skin Cancer Center of Lees Summit, Lee's Summit, Missouri
  - Saint Louis University, St Louis, Missouri
  - Somnos Clinical Research, Lincoln, Nebraska
  - Jubilee Clinical Research Inc, Las Vegas, Nevada
  - Excel Clinical Research, Las Vegas, Nevada
  - Las Vegas Clinical Trials, North Las Vegas, Nevada
  - Skin Cancer and Dermatology Institute, Reno, Nevada
  - Albuquerque Clinical Trials Incorporated, Albuquerque, New Mexico
  - Forest Hills Dermatology Group, Kew Gardens, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Sadick Research Group, New York, New York
  - OptiSkin Medical, New York, New York
  - Chear Center LLC, The Bronx, New York
  - DJL Clinical Research PLLC, Charlotte, North Carolina
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - Accellacare of Wilmington, Wilmington, North Carolina
  - The Skin Surgery Center for Clinical Research, Winston-Salem, North Carolina
  - Bexley Dermatology Research, Bexley, Ohio
  - Bernstein Clinical Research Center LLC, Cincinnati, Ohio
  - The Ohio State University, Gahanna, Ohio
  - Apex Clinical Research Center LLC, Mayfield Heights, Ohio
  - Dermatologist of Central States Clinical Research - Springfield, Springfield, Ohio
  - Unity Clinical Research, Oklahoma City, Oklahoma
  - Dermatology Research Center of Oklahoma, PLLC, Tulsa, Oklahoma
  - Essential Medical Research LLC, Tulsa, Oklahoma
  - Velocity Clinical Research Medford, Medford, Oregon
  - Oregon Medical Research Center, Portland, Oregon
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Best Skin Research, Camp Hill, Pennsylvania
  - Paddington Testing Company Inc, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Cumberland Skin Center, Hermitage, Tennessee
  - US Dermatology Partners Jollyville, Austin, Texas
  - Bellaire Dermatology Associates, Bellaire, Texas
  - US Dermatology Partners Cedar Park, Cedar Park, Texas
  - Driscoll Childrens Hospital, Corpus Christi, Texas
  - Alina Clinical Trials, LLC, Dallas, Texas
  - Dermatology Treatment and Research Center PA, Dallas, Texas
  - Zenos Clinical Research, Dallas, Texas
  - Texas Dermatology Research Center, Dallas, Texas
  - Newco 3A Research LLC, El Paso, Texas
  - Center For Clinical Studies PLLC, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Sante Clinical Research, Kerrville, Texas
  - Long and Harris Dermatology, Lubbock, Texas
  - Sms Clinical Research Limited Liability Company, Mesquite, Texas
  - Stride Clinical Research LLC, Missouri City, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Stryde Research Epiphany Dermatology, Southlake, Texas
  - The Woodlands Dermatology Associates, The Woodlands, Texas
  - Tanner Clinic, Murray, Utah
  - University of Utah MidValley Dermatology, Murray, Utah
  - Education and Research Foundation Inc, Forest, Virginia
  - Virginia Dermatology and Skin Cancer Center, Norfolk, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - MultiCare Institute for Research and Innovation, Spokane, Washington
- Argentina (14):
  - Conexa Investigacion Clinica SA, CABA, Buenos Aires
  - Cinme - Centro de Investigaciones Metabolicas, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Fundacion Respirar, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Universitario Austral, Derqui, Pilar, Buenos Aires
  - Framingham Centro Medico, La Plata, Buenos Aires
  - Buenos Aires Skin SA, Buenos Aires, Distrito Federal
  - Fundacion Cidea, Buenos Aires, Distrito Federal
  - Care- Centro de Alergia y Enfermedades Respiratorias, Buenos Aires, Distrito Federal
  - Instituto de Neumonologia y Dermatologia, Buenos Aires, Distrito Federal
  - Psoriahue Medicina Interdisciplinaria SRL, Buenos Aires, Distrito Federal
  - InAER - Investigaciones en Alergia y Enfermedades Respiratorias, CABA, Distrito Federal
  - Centro de Investigaciones Clinicas Instituto Especialidades De La Salud De Rosario, Rosario, Santa Fe Province
  - Fundacion Estudios Clinicos, Rosario, Santa Fe Province
  - Instituto de Diagnostico abc, Rosario, Santa Fe Province
- Australia (14):
  - Premier Specialists, Kogarah, New South Wales
  - St George Dermatology and Skin Cancer Centre, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - The Skin Centre, Benowa, Queensland
  - Princess Alexandra Hospital, South Brisbane, Queensland
  - Veracity Clinical Research, Woolloongabba, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - Emeritus Research Camberwell, Camberwell, Victoria
  - Skin Health Institute, Carlton, Victoria
  - Monash Childrens Hospital, Clayton, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Institute for Skin Health and Immunity, Mitcham, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- Austria (2):
  - Medizinische Universitaet Graz, Graz
  - Landeskrankenhaus Salzburg, Salzburg
- Belgium (7):
  - Universite Catholique de Louvain Cliniques Universitaires Saint Luc, Brussels
  - Grand Hopital de Charleroi - Site des Viviers, Charleroi
  - Universitair Ziekenhuis Gent, Ghent
  - Clinique Andre Renard, Herstal
  - Dermatologie Handelskaai, Kortrijk
  - Centre Hospitalier Universitaire de Liege - Sart Tilman, Liège
  - Dermatologie Maldegem, Maldegem
- Brazil (19):
  - Centro do Diagnostico e Pesquisa da Osteoporose do Espirito Santo, Vitória, Espírito Santo
  - Clinica Instituto Bahiano de Imunoterapia - Medicina, Reumatologia e Dermatologia ltda, Salvador, Estado de Bahia
  - Centro de Pesquisa Clínica da Universidade de Belo Horizonte - Unibh, Belo Horizonte, Minas Gerais
  - Ceti Centro Est Terap Inovadoras, Curitiba, Paraná
  - Universidade Federal do Parana, Curitiba, Paraná
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Ernesto Dornelles, Porto Alegre, Rio Grande do Sul
  - Alergoalfa Nucleo Diagnostico Tratamento e Pesquisa Clinica em Alergia, Barueri, São Paulo
  - Cecip Centro Est Clin Int Paulista, Jaú, São Paulo
  - Fundacao Abc - Centro Univ Fmabc, Santo André, São Paulo
  - Cemec Centro Multidisciplinar Estudos Clinicos, São Bernardo do Campo, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Ispem - Instituto Sao Jose dos Campos em Pesquisas Medicas, São José dos Campos, São Paulo
  - Instituto Pesquisa e Ensino em Saúde Infantil, São Paulo, São Paulo
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, São Paulo, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo
  - Consultoria Medica e Pesquisa Clinica Cmpc, Sorocaba, São Paulo
  - IBPClin Instituto Brasil de Pesquisa Clinica, Rio de Janeiro
- Bulgaria (5):
  - Medical Center Asklepii OOD, Dupnitsa
  - Medical Center Medconsult Pleven OOD, Pleven
  - Medical Center Excelsior OOD, Sofia
  - Diagnostic-Consultative Center Alexandrovska EOOD, Sofia
  - Diagnostic-Consultative Center - Fokus-5 - Medical Institution for Outpatient Care OOD, Sofia
- Canada (50):
  - Dermatology Research Institute Incorporated, Calgary, Alberta
  - Beacon Dermatology, Calgary, Alberta
  - Rejuvenation Dermatology Laser Calgary North, Calgary, Alberta
  - Laser Rejuvenation Clinics Edmonton D T Incorporated, Edmonton, Alberta
  - Stratica Dermatology, Edmonton, Alberta
  - Alberta Derma Surgery Centre, Edmonton, Alberta
  - Vida Clinical Research, Edmonton, Alberta
  - Skin Physicians Dermatology, Edmonton, Alberta
  - Interior Dermatology Centre, Kelowna, British Columbia
  - Doctor Chih-Ho Hong Medical Incorporated, Surrey, British Columbia
  - Enverus Medical Research, Surrey, British Columbia
  - Winnipeg Clinic Dermatology Research, Winnipeg, Manitoba
  - Wiseman Dermatology Research Incorporated, Winnipeg, Manitoba
  - Karma Clinical Trials, St. John's, Newfoundland and Labrador
  - CCA Medical Research Corp, Ajax, Ontario
  - SimcoDerm Medical and Surgical Dermatology Centre, Barrie, Ontario
  - Halton Pediatric Allergy, Burlington, Ontario
  - SKiN Health, Coburg, Ontario
  - Kingsway Clinical Research, Etobicoke, Ontario
  - Guelph Dermatology Research, Guelph, Ontario
  - LEADER Research, Hamilton, Ontario
  - Triple A Lab, Hamilton, Ontario
  - Centricity Research London Victoria, London, Ontario
  - Lynderm Research Inc, Markham, Ontario
  - DermEdge Research Incorporated, Mississauga, Ontario
  - Ryan Clinical Research Incorporated, Newmarket, Ontario
  - Allergy Research Canada Incorporated, Niagara Falls, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - Canadian Dermatology Centre, North York, Ontario
  - The Centre for Clinical Trials Inc, Oakville, Ontario
  - JRB Research Incorporated, Ottawa, Ontario
  - Dermatology Ottawa Research Centre, Ottawa, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - York Dermatology Clinic and Research Centre, Richmond Hill, Ontario
  - Oak Ridges Aesthetics Centre, Richmond Hill, Ontario
  - North York Research Incorporated, Toronto, Ontario
  - Toronto Research Centre Inc, Toronto, Ontario
  - FACET Dermatology, Toronto, Ontario
  - Research Toronto, Toronto, Ontario
  - Evidence Based Medical Educator Inc, Toronto, Ontario
  - Alliance Clinical Trials, Waterloo, Ontario
  - XLR8 Medical Research, Incorporated, Windsor, Ontario
  - Clinique de Dermatologie Rosemont, Montreal, Quebec
  - Innovaderm Research Inc, Montreal, Quebec
  - Recherche Clinique Sigma Incorporated, Québec, Quebec
  - Centre de Recherche Dermatologique du Quebec Metropolitain, Québec, Quebec
  - Clinique Medicale Saint Louis, Québec, Quebec
  - Skinsense Medical Research, Saskatoon, Saskatchewan
  - Saskatoon Dermatology Centre, Saskatoon, Saskatchewan
- Chile (5):
  - Hospital Base San Jose de Osorno, Osorno
  - Centro Medico Skinmed Spa, Santiago
  - Clinica Dermacross SA, Santiago
  - Fundacion Innovacion Cardiovascular Clinica Ensenada, Santiago
  - Centro Internacional de Estudios Clinicos, Santiago
- China (33):
  - Peking University Peoples Hospital, Beijing, Beijing Municipality
  - Beijing Childrens Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Childrens Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital Sun-Yat Sen University, Guangzhou, Guangdong
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital Sun Yat-sen University, Guangzhou, Guangdong
  - The Fist Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Shenzhen Childrens Hospital, Shenzhen, Guangdong
  - The First Hospital Of Hebei Medical University, Shijiazhuang, Hebei
  - Nanyang First Peoples Hospital, Nanyang, Henan
  - Sanmenxia Central Hospital, Sanmenxia, Henan
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Childrens Hospital, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Wuxi Second Peoples Hospital, Wuxi, Jiangsu
  - Wuxi Peoples Hospital, Wuxi, Jiangsu
  - Dermatology Hospital of Jiangxi Province, Nanchang, Jiangxi
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - Chengdu Second Peoples Hospital, Chengdu, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - Kunming Childrens Hospital, Kunming, Yunnan
  - Zhejiang Provincial Peoples Hospital, Hangzhou, Zhejiang
  - Affiliated Hangzhou First Peoples Hospital School of Medicine Westlake University, Hangzhou, Zhejiang
  - Ningbo NO 2 Hospital, Ningbo, Zhejiang
  - The First Affiliation Hospital Of Ningbo University, Ningbo, Zhejiang
  - Taizhou Central Hospital, Taizhou, Zhejiang
- Croatia (3):
  - Special Hospital for Medical Rehabilitation Naftalan, Ivanić-Grad
  - Children s Hospital Zagreb, Zagreb
  - University Hospital Centre Zagreb, Zagreb
- Czechia (14):
  - Kozni ambulance Kutna Hora sro, Kutná Hora
  - Dermamedica, sro, Náchod
  - Nemocnice Novy Jicin as, Nový Jičín
  - CCR Ostrava sro, Ostrava
  - Pratia Pardubice as, Pardubice
  - Fakultni nemocnice Plzen, Pilsen
  - Clintrial sro, Prague
  - Dermamedest sro, Prague
  - Pratia Prague sro, Prague
  - Kozni ambulance Fialova sro, Prague
  - Fakultni nemocnice Bulovka, Prague
  - Praglandia sro, Praha 5 - Smichov
  - Dermatologicka ambulance MUDr Petr Trestik, Svitavy
  - Krajska zdravotni as - Masarykova nemocnice Usti nad Labem oz, Ústí nad Labem
- Gentofte Hospital, Hellerup, Denmark
- Estonia (2):
  - North Estonia Medical Centre, Tallinn
  - Clinical Research Centre, Tartu
- Finland (3):
  - Clinical Research Services Helsinki, Helsinki
  - Oulun Yliopistollinen sairaala, Oulu
  - Terveystalo Tampere, Tampere
- France (10):
  - Hopital Prive d Antony, Antony
  - Polyclinique de Courlancy, Bezannes
  - Centre Hospitalier Regional Universitaire de Brest - Hopital Morvan, Brest
  - Centre Hospitalier Regional Universitaire de Lille - Hopital Claude Huriez, Lille
  - Centre Hospitalier de Bretagne Sud - Hopital du Scorff, Lorient
  - Cabinet du Docteur Ruer-Mulard Mireille, Martigues
  - Centre Hospitalier Universitaire Archet 2, Nice
  - Hopital Saint Louis, Paris
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
  - Centre Hospitalier Universitaire de Rouen - Hopital Charles Nicolle, Rouen
- Germany (25):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Charite - Universitaetsmedizin Berlin, Campus Mitte, Berlin
  - Clinical Research Services Berlin GmbH, Berlin
  - Hautarztpraxis Dr Niesmann und Dr Othlinghaus, Bochum
  - Rosenpark Research GmbH, Darmstadt
  - Universitaetsklinikum Dresden, Dresden
  - Universitaetsklinikum Frankfurt, Frankfurt am Main
  - Universitaetsmedizin Goettingen - Georg-August-Universitaet, Göttingen
  - Institute for Health Services Research in Dermatology and Nursing, Hamburg
  - Hautaerzte Zentrum Hannover, Hanover
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Schleswig-Holstein - Kiel, Kiel
  - Velocity Clinical Research, Leipzig
  - Dermatologische Gemeinschaftspraxis-Mahlow, Mahlow
  - Universitaetsmedizin Mainz, Mainz
  - Beldio Research GmbH, Memmingen
  - Hautmedizin Saar, Merzing
  - Klinikum rechts der Isar der TUM, München
  - Universitaetsklinikum Muenster, Münster
  - KliFOs Klinische Forschung Osnabrueck, Osnabrück
  - Hautarztpraxis Mortazawi, Remscheid
  - Hautarztpraxis Dres Leitz und Kollegen, Stuttgart
  - Universitaetsklinikum Tuebingen, Tübingen
  - Helios Klinikum Wuppertal, Wuppertal
  - CentroDerm GmbH, Wuppertal
- Greece (7):
  - University General Hospital Attikon, Athens
  - Andreas Syngros Hospital Of Venereal And Dermatological Diseases, Athens
  - University General Hospital of Ioannina, Ioannina
  - General University Hospital of Larissa, Larissa
  - General Hospital Of Nea Ionia Konstantopouleio Patision, Nea Ionia
  - Geniko Nosokomeio Peiraia Tzaneio, Piraeus
  - Papageorgiou General Hospital, Thessaloniki
- Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong
- Hungary (11):
  - Trial Pharma Kft, Békéscsaba
  - Csalogany Orvosi Kozpont, Budapest
  - Clinexpert Kft, Budapest
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Gyongyosi Bugat Pal Korhaz, Gyöngyös
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz, Kaposvár
  - DermaMed Research Kft, Orosháza
  - Allergo-Derm Bakos Kft, Szolnok
  - Medmare Bt, Veszprém
  - Obudai Egeszsegugyi Centrum Kft, Zalaegerszeg
- Sheba Medical Center, Ramat Gan, Israel
- Italy (8):
  - Universita degli Studi Gabriele D Annunzio di Chieti e Pescara, Chieti
  - Ospedale San Salvatore, LAquila
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli, Napoli
  - Azienda Ospedaliera di Perugia Ospedale Santa Maria della Misericordia, Perugia
  - Azienda Ospedaliera Policlinico Umberto I, Roma
  - IRCCS Istituto Clinico Humanitas, Rozzano MI
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino, Torino
- Japan (51):
  - Aichi Medical University Hospital, Nagakute-shi, Aichi-ken
  - Fukui Dermatology Clinic, Nagoya, Aichi-ken
  - Japan Community Healthcare Organization Chukyo Hospital, Nagoya, Aichi-ken
  - Central Clinic, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Miyata Dermatology Clinic, Matsudo-shi, Chiba
  - International University of Health and Welfare Narita Hospital, Narita-shi, Chiba
  - Ekihigashi Dermatology Allergy Clinic, Fukuoka, Fukuoka
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Matsuo Clinic, Fukuoka, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Asahikawa City Hospital, Asahikawa-shi, Hokkaido
  - Takagi Dermatological Clinic, Obihiro-shi, Hokkaido
  - Medical Corporation Kojinkai Sapporo Skin Clinic, Sapporo, Hokkaido
  - Yoshimura Child Clinic, Akashi-shi, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - Tokyo Medical University Ibaraki Medical Center, Inashiki-gun, Ibaraki
  - Kaji Dermatology Clinic, Nonoichi-shi, Ishikawa-ken
  - Iwate Medical University Uchimaru Medical Center, Morioka, Iwate
  - Takeoka Dermatology Clinic, Marugame-shi, Kagawa-ken
  - Katahira Dermatology Urology Clinic, Kagoshima, Kagoshima-ken
  - Kosugi Dermatology Clinic, Kawasaki-shi, Kanagawa
  - Nippon Medical School Musashikosugi Hospital, Kawasaki-shi, Kanagawa
  - St Marianna University Hospital, Kawasaki-shi, Kanagawa
  - National Hospital Organization Sagamihara National Hospital, Sagamihara-shi, Kanagawa
  - Nomura Dermatology Clinic, Yokohama, Kanagawa
  - Showa Medical University Northern Yokohama Hospital, Yokohama, Kanagawa
  - Yokohama City Minato Red Cross Hospital, Yokohama, Kanagawa
  - Jouzan Hihuka Hinyoukika Clinic, Kumamoto, Kumamoto
  - Suizenji Dermatology Clinic, Kumamoto, Kumamoto
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Rakuwakai Otowa Hospital, Kyoto, Kyoto
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Osaka Habikino Medical Center, Habikino-shi, Osaka
  - Mochida Dermatology Clinic, Izumiotsu-shi, Osaka
  - Yoshioka Dermatology Clinic, Neyagawa, Osaka
  - Dermatology and Ophthalmology Kume Clinic, Sakai-shi, Osaka
  - JA Shizuoka Kohseiren Enshu Hospital, Hamamatsu, Shizuoka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Dokkyo Medical University Hospital, Shimotsuga-gun, Tochigi
  - Mildix Skin Clinic, Adachi-ku, Tokyo
  - Teikyo University Hospital, Itabashi-ku, Tokyo
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
  - Mita Dermatology Clinic, Minato-ku, Tokyo
  - Naoko Dermatology Clinic, Setagaya-ku, Tokyo
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo
  - Showa Medical University Hospital, Shinagawa-ku, Tokyo
  - Seibo International Catholic Hospital, Shinjuku-ku, Tokyo
  - Yamate Dermatology Clinic, Shinjuku-ku, Tokyo
  - Sugamo Kobayashi Derma Clinic, Toshima-ku, Tokyo
  - Shirasaki Dermatology Clinic, Takaoka-shi, Toyama
- Latvia (3):
  - Outpatient clinic Veselibas Centrs 4, Riga
  - Outpatient clinic Veselibascentrs 4, Riga
  - Smite Aija practice in dermatology and venerology, Talsi
- Malaysia (4):
  - Hospital Sultan Ismail, Johor Bahru, Johor
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Hospital Pulau Pinang, George Town, Pulau Pinang
- Mexico (2):
  - Clínica de Enfermedades Crónicas y de Procedimientos Especiales, Morelia, Michoacán
  - Phylasis Clinical Research, Cuautitlán Izcalli
- Netherlands (3):
  - Bravis Ziekenhuis, Bergen op Zoom
  - Universitair Medisch Centrum Groningen, Groningen
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (27):
  - ClinicMed Daniluk Nowak Spolka komandytowa, Bialystok
  - Dermapolis Medical Dermatology Center dr n med Edyta Gebska, Chorzów
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - AKK Medical Spolka z ograniczona odpowiedzialnoscia Centrum Medyczne Tu sie leczy, Gdansk
  - GynCentrum Spzoo NZOZ Holsamed - Oddzial Libero, Katowice
  - Centrum Medyczne Angelius Provita, Katowice
  - Specjalistyczny Gabinet Dermatologiczny Aplikacyjno-Badawczy Marek Brzewski Pawel Brzewski SpCywilna, Krakow
  - Diamond Clinic Spolka z Ograniczona Odpowiedzialnoscia Diamond Medical Center, Krakow
  - Centrum Terapii Wspolczesnej J M Jasnorzewska Spolka Komandytowo Akcyjna, Lodz
  - AppleTreeClinics Network Spzoo, Lodz
  - Ip Clinic Sp zoo, Lodz
  - Amicare Spolka z ograniczona odpowiedzialnoscia Spolka Komandytowa Amicare Centrum Medyczne, Lodz
  - Clinical Best Solutions Sp zoo Spolka Komandytowa, Lublin
  - Centrum Zdrowia i Urody Maxxmed, Lublin
  - Centrum Badawcze Panaceum Agnieszka Brzezicka Magdalena Lenkiewicz Spzoo, Malbork
  - Twoja przychodnia Ncm, Nowa Sól
  - Twoja przychodnia Pcm, Poznan
  - Centrum Zdrowia Dziecka i Rodziny Im Jana Pawla II w Sosnowcu Osrodek Badan Klinicznych, Sosnowiec
  - Twoja Przychodnia Scm, Szczecin
  - Alergo-Med Osrodek Badan Klinicznych sp zoo, Tarnów
  - Klinika Osipowicz and Turkowski Sp zoo, Warsaw
  - High Med Przychodnia Specjalistyczna, Warsaw
  - Evimed sp zoo centrum medyczne evimed, Warsaw
  - Klinika Ambroziak Dermatologia, Warsaw
  - Royalderm Agnieszka Nawrocka, Warsaw
  - DermMedica Spzoo Centrum Columbus, Wroclaw
  - Dermaceum Spolka z Ograniczona Odpowiedzialnoscia Dermaceum Centrum Medyczne, Wroclaw
- Portugal (5):
  - Unidade de Saude Local de Almada-Seixal, EPE - Hospital Garcia de Orta, Almada
  - Unidade Local de Saude de Coimbra, EPE, Coimbra
  - Hospital Cuf Descobertas, Lisbon
  - Unidade Local de Saude de Santo Antonio, EPE - Hospital de Santo Antonio, Porto
  - Unidade Local de Saude de Sao Joao, EPE - Hospital de Sao Joao, Porto
- Gcm Medical Group, Psc, San Juan, Puerto Rico
- Derma Cluj, Cluj-Napoca, Romania
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - National Skin Centre, Singapore
- Slovakia (6):
  - Fakultna Nemocnica s poliklinikou F D Roosevelta Banska Bystrica, Banská Bystrica
  - Maxderm, sro, Bardejov
  - Univerzitna nemocnica Bratislava - Nemocnica Stare Mesto, Bratislava
  - Derma therapy, spol s ro, Bratislava
  - Sanare spol sro, Svidník
  - Kaderma Majtan, sro, Topoľčany
- Slovenia (2):
  - Univerzitetni klinicni center Ljubljana, Ljubljana
  - Univerzitetni Klinicni Center Maribor, Maribor
- Hiway Medical Centre, Westville, Durban, KwaZulu-Natal, South Africa
- South Korea (19):
  - Korea University Ansan Hospital, Ansansi, Gyeonggido
  - SoonChunHyang University Hospital Bucheon, Bucheon-si, Gyeonggi-do
  - Chosun University Hospital, Gwangju
  - The Catholic University of Korea Incheon St Marys Hospital, Incheon
  - Inha University Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - National Medical Center, Seoul
  - Konkuk University Medical Center, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Ewha Womans University Seoul Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Ajou University Hospital, Suwon-si, Gyeonggi-do
- Spain (20):
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Universitario Virgen Macarena, Seville, Andalusia
  - Hospital Universitario Basurto, Bilbao, Basque Country
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Universitari Germans Trias i Pujol, Badalona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Catalonia
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, Galicia
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital General Universitario de Alicante, Alicante, Valencia
  - Hospital de Manises, Manises, Valencia
  - Hospital Arnau de Vilanova de Valencia, Valencia, Valencia
  - Hospital Universitario de La Princesa, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Miguel Servet, Zaragoza
- Switzerland (3):
  - Inselspital Bern, Bern
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Universitaetsspital Zuerich, Zurich
- Taiwan (6):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital Taipei Branch, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Thailand (4):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Thammasat University Hospital, Pathum Thani
- Turkey (Türkiye) (9):
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Gaziantep Universitesi Tip Fakultesi Hastanesi, Gaziantep
  - Istanbul Universitesi Istanbul Tip Fakultesi Hastanesi, Istanbul
  - Acibadem Altunizade Hastanesi, Istanbul
  - Marmara Universitesi Tip Fakultesi Hastanesi, Istanbul
  - Bakircay Universitesi Cigli Egitim ve Arastirma Hastanesi, Izmir
  - Erciyes Universitesi Tip Fakultesi Hastanesi, Kayseri
  - Kocaeli Universitesi Tip Fakultesi Hastanesi, Kocaeli
  - Ondokuz Mayis Universitesi Tip Fakultesi Hastanesi, Samsun
- United Kingdom (6):
  - Alder Hey Childrens Hospital, Liverpool
  - Whipps Cross University Hospital, London
  - The Royal Free Hospital, London
  - Guys Hospital, London
  - Salford Care Organisation, Salford
  - Accellacare Yorkshire, Shipley

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Guttman-Yassky E, Simpson E, Bissonnette R, Eichenfield LF, Kabashima K, Luna PC, Hercogova JT, Spelman L, Worm M, Esfandiari E, Arai T, Mano H, Charuworn P, Wang A, Kricorian G. ROCKET: a phase 3 program evaluating the efficacy and safety of rocatinlimab in moderate-to-severe atopic dermatitis. Immunotherapy. 2025 Feb;17(2):83-94. doi: 10.1080/1750743X.2025.2464528. Epub 2025 Feb 26. PMID 40012373
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com